CLINICAL TRIAL: NCT00319228
Title: A Phase II/III Pivotal Trial Evaluating the Safety, Pharmacokinetic Properties and Efficacy of a Plasma-Derived Anti-thrombin III Concentrate With Administration in Surgery, Pregnancy and Thromboembolic or Thrombotic Events
Brief Title: Safety, Pharmacokinetics and Efficacy of an ATIII Concentrate
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Grifols Biologicals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IG-401
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Antithrombin III Deficiency
Keywords: AT-III deficiency; AT-III concentrate; Bleeding disorders; Blood disorders
MeSH Terms: conditions — Antithrombin III Deficiency; Hemostatic Disorders; Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Antithrombin III (Experimental)
  Interventions: Drug: Plasma-derived AT-III concentrate

INTERVENTIONS:
Drug: Plasma-derived AT-III concentrate — Segment I: A single dose IV infusion of 50 IU/kg of ATIII-DAF/DI will be administered to each patient.
  Segment II: A single dose or multiple doses depending on the subject's ATIII plasma levels and patient's specific treatment plan.

SUMMARY:
To assess the safety, pharmacokinetics and efficacy of a plasma-derived AT-III concentrate in the treatment of subjects with congenital AT-III deficiency.

DETAILED DESCRIPTION:
This study will be a prospective, unblinded, non-randomized, open-label, multi-center Phase II/III study with 2 segments, i.e. a PK evaluation (Segment I), and an assessment of prophylaxis in surgical interventions and pregnancy/delivery, (Segment II). During the PK segment (Segment I), the subjects would remain on their current anticoagulation therapy except for subjects on heparin therapy where a wash-out period of at least 5 half-lives would be required. In total, 15 subjects with congenital ATIII Deficiency will be enrolled for the PK assessment (Segment I).

For Segment II, fifteen episodes will be treated. Recruitment of individual subjects with high risk for venous thrombosis for Segment II of this study is necessary because of the rarity of Antithrombin deficiency in the population.

ELIGIBILITY:
Inclusion Criteria:

* Congenital ATIII deficiency documented by determination of plasma levels of ATIII off all therapies. Specifically, the baseline levels of ATIII activity should be equal to or less than 60%.
* Age >12 years with a body weight of no less than 30 kg.
* Have not participated in another investigational study for at least 30 days. For Segment II, enrollment requires a pregnancy/delivery or a surgical procedure (it should be a major surgery although data from a minor surgery will also be collected).
* Documented personal history of major thromboembolic or thrombotic event.
* Male or female
* HIV, HBV, HCV, HAV and PARVO B19 status known prior to entry.
* The subject is willing to comply with all aspects of the protocol, including blood sampling, for the duration of the study.
* The subject has signed an informed consent form (if at least 18 years old), or the subject's parent or legal guardian has signed the informed consent form. Subjects below the age of 18 years will also be asked to sign an assent form. All consent and assent forms must be approved in advance by the Institutional Review Board of the investigator's institution.
* Patients with heparin-associated thrombocytopenia who require anticoagulation with non-heparin containing drugs will be eligible if they can be safely transitioned during the washout period for the Segment I PK study.
* If pregnant, a woman must be Parvo B19 IgG antibody positive.

Exclusion Criteria:

* Acquired deficiency of ATIII.
* Receiving concomitant treatment for thrombophilic disorders other than ATIII deficiency.
* Inability or unwillingness to comply with the protocol requirements.
* History of anaphylactic reaction(s) to blood or blood components.
* Allergies to excipients.
* Liver function tests >/= 2.5 X ULN
* Serum creatinine >1.2 X ULN.
* Urine >/= 2+ protein with urine dipstick test.
* The subject is known to have abused alcohol or illicit drugs within the past 12 months.
* The subject is unlikely to adhere to the protocol requirements of the study or is likely to be uncooperative or unable to provide a storage serum sample at the screening visit.
* Patients on heparin-treatment who, for clinical reasons, cannot safely be discontinued from heparin therapy during the PK segment.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
The primary objectives of this clinical study are to: | 2 years
Assess the pharmacokinetic (PK) profile of AT-III in congenital AT-III deficient patients | 1 year
To measure the in vivo recovery and half-life of AT-III. | 1 year
To assess the clinical safety and tolerability of AT-III-DAF/DI. | 1 year

SECONDARY OUTCOMES:
To assess clinical efficacy by preventing thromboembolic or thrombotic events (prophylaxis) in individuals with congenital AT-III deficiency who are undergoing surgical procedures or who are pregnant and undergoing parturition. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Paul Pinciaro, PhD, Study Director — Grifols Biologicals, LLC